CLINICAL TRIAL: NCT07377149
Title: Quality Improvement Intervention on Utilization of Arterial Grafts for Coronary Artery Bypass Grafting
Brief Title: Improving the Quality of Coronary Artery Bypass Grafting
Acronym: CABG Quality
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Collaborators: Chinese Academy of Medical Sciences, Fuwai Hospital (Other); Shandong Provincial Hospital (Other Government); The First Affiliated Hospital with Nanjing Medical University (Other); Guangdong Provincial People's Hospital (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); West China Hospital (Other); First Affiliated Hospital of Wenzhou Medical University (Other); Ruijin Hospital (Other); The General Hospital of Northern Theater Command (Other); Central China Fuwai Hospital of Zhengzhou University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2025-2849; 2025ZD0546704 (Other: Noncommunicable Chronic Diseases-National Science and Technology Major Project)
Record Dates: First submitted 2025-12-23; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Coronary Artery Bypass Grafting (CABG)
Keywords: coronary artery bypass grafting; quality improvement; arterial graft
MeSH Terms: interventions — Methods; Health Personnel; Hospitals

STUDY DESIGN:
Intervention Model Description: This is a stepped-wedge cluster randomized trial (SW-CRT) with a self-controlled design. Hospitals were categorized into two groups based on their internal mammary artery graft usage rates (low or high), forming two SW-CRT.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Improving the utilization rate of arterial grafts for coronary artery bypass grafting (Other): In this stepped-wedge cluster randomized trial (SW-CRT) with a self-controlled design, hospitals were categorized into two groups according to their internal mammary artery graft usage rates, thereby forming two SW-CRT. Healthcare professionals at these hospitals will receive tailored interventions. The effectiveness of each intervention is assessed by comparing the usage rates before and after implementation within each SW-CRT.
  Interventions: Behavioral: Interventions for healthcare professionals in hospitals with low usage rates; Behavioral: Interventions for healthcare professionals in hospitals with high usage rates

INTERVENTIONS:
Behavioral: Interventions for healthcare professionals in hospitals with low usage rates — Hospitals with low usage rates aim to improve internal mammary artery graft utilization through interventions including education, theoretical training, technical training, conference exchanges, and regular feedback on quality monitoring results.
Behavioral: Interventions for healthcare professionals in hospitals with high usage rates — Hospitals with already high usage rates focus on increasing multi-arterial graft usage rates through similar intervention methods such as education, theoretical training, technical training, conference exchanges focus on multi-arterial graft use. The usage rates of multi-arterial graft for each hospital will be regular feed backed.

SUMMARY:
This is a healthcare quality improvement study focused on increasing the utilization of arterial grafts in isolated coronary artery bypass grafting (CABG). Evidence indicates that arterial grafts, compared with venous grafts, provide superior long-term patency, which are recommended to use by the clinical practice guidelines.

In hospitals where the use of the internal mammary artery as a graft is relatively low(<90%) among CABG patients, multiple interventions will be implemented to improve its adoption rate.

In hospitals where internal mammary artery graft utilization is already high(≥90%), various interventions will be introduced to promote the use of multiple arterial grafts (defined as the use of two or more arterial conduits).

The study targets healthcare professionals as the primary subjects of intervention, with no direct interventions applied to patients during the study period. Changes in the internal mammary artery graft utilization rate and the multiple arterial graft utilization rate before and after the intervention will serve as the primary endpoints for evaluating intervention effectiveness in the two types of hospitals, respectively.

ELIGIBILITY:
Patients whose data used to monitor the quality

Inclusion Criteria:

Aged ≥ 18 years old； Indicated for CABG and undergoing CABG.

Exclusion Criteria:

History of prior CABG; Concurrent other cardiac surgeries on the day of CABG; Malignant tumor or life expectancy < 1 year;

* 50% stenosis of left subclavian artery; Pregnant women; Individuals diagnosed with mental illness or cognitive impairment (International Classification of Diseases-10 codes F01-F99); Patients considered by the investigator to have other factors unsuitable for inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8700 (Estimated)
Dates: Start 2026-03-15 (Estimated); Primary Completion 2029-01 (Estimated); Study Completion 2029-07 (Estimated)

PRIMARY OUTCOMES:
Hospitals with low usage rates of internal mammary artery: internal mammary artery graft utilization rate | Duration of hospital stay(from date of admission to date of discharge)
  Internal mammary artery graft utilization rate: the utilization rate of at least one internal mammary artery graft in patients received isolated coronary artery bypass grafting.
Hospitals with high usage rates of internal mammary artery: multiple arterial graft utilization rate | Duration of hospital stay(from date of admission to date of discharge)
  Multiple arterial graft utilization rate: the utilization rate of two or more arterial conduits in patients received isolated coronary artery bypass grafting.

SECONDARY OUTCOMES:
In-hospital all-cause mortality rate | Duration of hospital stay(from date of admission to date of discharge)
  The in-hospital all-cause mortality rate of patients received isolated coronary artery bypass grafting.

IPD SHARING:
Plan to Share IPD: No